CLINICAL TRIAL: NCT06035068
Title: Sentinel Lymph Node Mapping and Detection With Indocyanine Green and Spy-Phi Handheld Camera Technology in Early-Stage Vulvar Cancer (PILOT)
Brief Title: SLN Mapping and ICG Dye for Vulvar Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00004163
Record Dates: First submitted 2023-09-06; First posted 2023-09-13 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Vulva Cancer
MeSH Terms: conditions — Vulvar Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Combined ICG dye and blue tracer dye: This study is being done to see if a different way of finding and removing lymph nodes during surgery, using a special camera and a dye called Indocyanine Green (ICG), works as well as the usual method with blue dye plus a radioactive tracer called radiocolloid. By comparing the two ways directly, we hope to make it simpler for people with vulvar cancer to get their lymph nodes checked during surgery.
  Interventions: Drug: Indocyanine green

INTERVENTIONS:
Drug: Indocyanine green — Indocyanine green (ICG) is a fluorescent dye that has been used for the imaging of cancers in the body for more than 30 years.
  Other Names: ICG dye

SUMMARY:
Doctors typically use blue dye to assist in locating and extracting lymph nodes for biopsy. However, this process can prove somewhat challenging for both patients and medical teams due to its need for extensive coordination and the assistance of a nuclear medicine team. Some studies have talked about using a different method to find these lymph nodes using a special dye called Indocyanine Green (ICG). This method involves shining a special camera on the skin. So far, no studies have directly compared the ICG method to the standard blue dye. The ICG camera could make things easier for patients and doctors, and more patients might choose to have their lymph nodes checked with this new method. The goal of our study is to see if using the ICG dye is just as good as the standard method of blue dye.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Patients with early-stage SCC (diameter <4 cm) of the vulva without suspicious lymph nodes at palpation or imaging who are planned for surgery at Tufts Medical Center.
* Patients with squamous cell carcinoma, depth of invasion > 1mm
* Patients with T1 or T2 tumors (FIGO staging) < 4 cm, not encroaching in urethra or anus with clinically negative inguinofemoral lymph nodes
* Localization and size of the tumor are such that perilesional injection of the tracers at three or four sites is possible
* Preoperative imaging do not show enlarged (<1.5 cm)/ suspicious nodes
* Willing and able to give informed consent

Exclusion Criteria:

* Inoperable tumors and tumors with diameter > 4 cm
* Patients with inguinofemoral lymph nodes that are palpable on clinical exam suspicious for metastases or with cytologically proven inguinofemoral lymph node metastases
* Radiologically enlarged (>1.5 cm) inguinofemoral lymph nodes
* Patients with multifocal tumors
* Pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 10 participants fitting the above criteria at Tufts Medical Center
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Detection Rate of SLNs using ICG Dye vs Blue Dye at Patient Level | Data collection at time of surgery
  * Report the detection rate of SLNs using ICG dye for sentinel lymph node mapping.
  * Report the detection rate of SLNs using blue dye for sentinel lymph node mapping.
  * Compare the two detection rates using a chi-squared test or Fisher's exact test, depending on the sample size.
Clustered Analysis at the Hemi-Pelvis Level | Data collection at time of surgery
  * Use generalized estimating equations (GEE) or mixed-effects logistic regression models to account for the clustering effect.
  * Include a random effect for each patient to address the correlation between SLNs within the same patient's hemi-pelvis.
  * Assess the significance of dye type using the Wald test or likelihood ratio test.
  * Report odds ratios, confidence intervals, and p-values for the effect of dye type on SLN detection.
3. Difference in SLNs Detected in Blue vs Green Dye when Data is Clustered at Hemi-Pelvis Level | Data collection at time of surgery
  * Report the proportion of SLNs detected using blue dye in each hemi-pelvis.
  * Report the proportion of SLNs detected using ICG dye in each hemi-pelvis.
  * Use a paired t-test or Mcnemar's test to compare the proportions within each hemi-pelvis.
  * Account for the clustering effect by using mixed-effects models

SECONDARY OUTCOMES:
Sensitivity, Specificity, and Negative Predictive Value of ICG Dye vs Standard Blue Dye | Data collection at time of surgery
  * Create a 2x2 contingency table for sensitivity, specificity, and negative predictive value.
  * Sensitivity = (True Positives) / (True Positives + False Negatives).
  * Specificity = (True Negatives) / (True Negatives + False Positives).
  * Negative Predictive Value = (True Negatives) / (True Negatives + False Negatives).

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Gonzalez, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Te Grootenhuis NC, van der Zee AG, van Doorn HC, van der Velden J, Vergote I, Zanagnolo V, Baldwin PJ, Gaarenstroom KN, van Dorst EB, Trum JW, Slangen BF, Runnebaum IB, Tamussino K, Hermans RH, Provencher DM, de Bock GH, de Hullu JA, Oonk MH. Sentinel nodes in vulvar cancer: Long-term follow-up of the GROningen INternational Study on Sentinel nodes in Vulvar cancer (GROINSS-V) I. Gynecol Oncol. 2016 Jan;140(1):8-14. doi: 10.1016/j.ygyno.2015.09.077. Epub 2015 Sep 30. PMID 26428940
- [Background] Covens A, Vella ET, Kennedy EB, Reade CJ, Jimenez W, Le T. Sentinel lymph node biopsy in vulvar cancer: Systematic review, meta-analysis and guideline recommendations. Gynecol Oncol. 2015 May;137(2):351-61. doi: 10.1016/j.ygyno.2015.02.014. Epub 2015 Feb 20. PMID 25703673
- [Background] Hutteman M, van der Vorst JR, Gaarenstroom KN, Peters AA, Mieog JS, Schaafsma BE, Lowik CW, Frangioni JV, van de Velde CJ, Vahrmeijer AL. Optimization of near-infrared fluorescent sentinel lymph node mapping for vulvar cancer. Am J Obstet Gynecol. 2012 Jan;206(1):89.e1-5. doi: 10.1016/j.ajog.2011.07.039. Epub 2011 Jul 30. PMID 21963099
- [Background] Crane LM, Themelis G, Arts HJ, Buddingh KT, Brouwers AH, Ntziachristos V, van Dam GM, van der Zee AG. Intraoperative near-infrared fluorescence imaging for sentinel lymph node detection in vulvar cancer: first clinical results. Gynecol Oncol. 2011 Feb;120(2):291-5. doi: 10.1016/j.ygyno.2010.10.009. Epub 2010 Nov 6. PMID 21056907